CLINICAL TRIAL: NCT02457884
Title: Effectiveness of Training in Reading Rehabilitation for Patients With Diabetic Macular Oedema (DMO)- Randomized Controlled Trial
Brief Title: Effectiveness of Training in Reading Rehabilitation for Patients With Diabetic Macular Oedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Allen MY Cheong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 12131601
Record Dates: First submitted 2015-05-25; First posted 2015-05-29 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Macular Oedema; Parafoveal Scotoma
Keywords: Diabetic macular oedema; Perceptual learning; Chinese; Hong Kong
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Temporal Group (Active Comparator): Receive 6 weekly 1-hour training sessions by Trigrams (A tailor made reading-task training programme).
  Interventions: Other: Temporal Group
- Spatial Group (Active Comparator): Receive 6 weekly 1-hour training sessions by Trigrams (A tailor made reading-task training programme).
  Interventions: Other: Spatial Group
- Combined Group (Active Comparator): Receive 6 weekly 1-hour training sessions by Trigrams (A tailor made reading-task training programme).
  Interventions: Other: Combined Group
- Control Group (Placebo Comparator): Receive 6 weekly 1-hour training sessions of leisure reading activities
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Temporal Group — Visual Processing Training
  Arms: Temporal Group
Other: Spatial Group — Spatial visual span training
  Arms: Spatial Group
Other: Combined Group — Visual processing speed and spatial visual span training
  Arms: Combined Group
Other: Control Group — Leisure reading activities
  Arms: Control Group

SUMMARY:
Diabetic macular oedema (DMO) is a sight-threatening problem for diabetic patient who has swelling in macula. Patients with DMO can receive laser treatment and achieve good acuity finally. However, some patients still have difficulties in reading even after proper treatment.

In this project, the investigators aimed to explore the effectiveness of different training paradigms in improving reading performance in patients with DMO.

DETAILED DESCRIPTION:
Patients with diabetic macular oedema (DMO), after receiving laser photocoagulation, achieved good outcomes in distance acuity. However, some patients, particularly those developing parafoveal scotoma, still had difficulty in reading. Inability to read or reading very slowly leads to the potential loss of job, as well as the enjoyment of reading for leisure.

In this study, the investigators aimed to investigate the effectiveness of reading rehabilitation using perceptual learning paradigms in enhancing reading performance in patients with reading difficulties due to DMO. Also, the fundamental mechanisms explaining the reading problems in patients with DMO reading Chinese will be examined.

The investigators hypothesize that the perceptual training would show an improvement in reading. The investigators' primary hypothesis is that temporal visual processing speed and spatial visual span will be improved after perceptual training. The investigators' secondary hypothesis is that the reading speed and fixation stability will be improved after training.

ELIGIBILITY:
Inclusion Criteria:

* Able to read Chinese.
* No formal vision rehabilitation training in reading after vision loss
* Diagnosis of diabetic macular oedema (DMO) and had previous treatment with laser and / or intravitreal injections
* Reasonable control of blood glucose level (HbA1c <10) to minimize the impact of vision fluctuation
* Education level of 6 years or more (primary school or above)

Exclusion Criteria:

* Receive any types of eye treatments other than those mentioned above
* Any diagnosed ocular diseases other than DMO
* Severe medical problems or self reported neurological or cognitive disorders
* Serious hearing impairment
* Previously attended vision rehabilitation clinic

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in visual processing speed | Change from baseline at week 6 and change from baseline at week 12 week
  Using trigrams to measure the character-recognition accuracy while characters are presented at different exposure times
Change in visual span size | Change from baseline at week 6 and change from baseline at week 12 week
  Using trigrams to measure the character-recognition accuracy while characters are presented at different positions

SECONDARY OUTCOMES:
Change in reading performance | Change from baseline at week 6 and change from baseline at week 12 week
  Measured in three different ways for Chinese:
  1. Rapid serial visual presentation (RSVP)
  2. Sentence reading (MNREAD)
  3. Passage reading (IReST)
Change in fixation stability | Change from baseline at week 6 and change from baseline at week 12 week
  Fixation stability will be measured by MP-1 microperimeter.
Change in Chinese version of Impact of Visually Impaired (C-IVI) measure | Change from baseline at week 6 and change from baseline at week 12 week
  Self evaluated instrument to measure vision related restriction of participation in daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Ming Yan Cheong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Allen MY Cheong, Hong Kong, China